CLINICAL TRIAL: NCT02890251
Title: Visual Maturation in Premature Newborns According to Factors Influencing Its Development
Acronym: PREMAVISION
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Professor, Central Hospital, Nancy, France
Other Study IDs: PSS2016/PREMAVISION-HASCOET/VS
Record Dates: First submitted 2016-08-18; First posted 2016-09-07 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Delayed Visual Maturation
Keywords: Infant; Premature; Diseases
MeSH Terms: conditions — Premature Birth; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose is to describe the level of visual maturation of premature newborns at term equivalent age.

The secondary purpose is to determine factors associated to an altered level of visual maturation, through an exploratory approach.

ELIGIBILITY:
Inclusion Criteria:

* Infants born before 33 weeks of amenorrhea and hospitalized at CHRU Nancy

Exclusion Criteria:

* Parental opposition
* Ocular malformation
* Face malformation
* Cranial stenosis
* Chromosomal abnormality

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature babies, born before 33 weeks of amenorrhea and hospitalized at CHRU Nancy, evaluated at term equivalent age.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2016-02-01; Primary Completion 2016-06-30 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Measurement of Visual Acuity by Baby Vision Cards | Baseline
  Baby Vision cards are the French equivalent of Teller Cards - The measurement will be done at the term equivalent age : at the inclusion

SECONDARY OUTCOMES:
Control of the Retina by Retinal Camera | Baseline
  Use of Retcam to diagnose Retinopathy of Prematurity - The measurement will be done at the term equivalent age : at the inclusion
Measurement of cycloplegic refraction by mydriaticum 0.5% | Baseline
  The measurement will be done at the term equivalent age : at the inclusion
Presence, absence of light reflex by clinical evaluation | Baseline
  The measurement will be done at the term equivalent age : at the inclusion
Presence, absence or abnormality of visual fixation by clinical observation | Baseline
  The measurement will be done at the term equivalent age : at the inclusion
Analysis of visual cortex with MRI | Baseline
  Determinants of indices of cerebral volume in former very premature infants and their relation to visual maturation. The measurement will be done at the term equivalent age : at the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel HASCOET, Pr, Principal Investigator — Maternité Régionale Universitaire A. Pinard CHRU Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wirth M, Naud A, Schmitt E, Clerc-Urmes I, Hascoet JM. Visual Maturation at Term Equivalent Age in Very Premature Infants According to Factors Influencing Its Development. Front Physiol. 2018 Nov 20;9:1649. doi: 10.3389/fphys.2018.01649. eCollection 2018. PMID 30515105